CLINICAL TRIAL: NCT02482142
Title: The Role of Phosphorus in Diet Induced Thermogenesis of Both Lean and Obese Subjects
Brief Title: The Role of Phosphorus in Diet Induced Thermogenesis (DIT) of Both Lean and Obese Subjects
Acronym: PinDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NUT.OO.22
Record Dates: First submitted 2015-03-25; First posted 2015-06-26 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: phosphorus; lean; obese; energy expenditure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- phosphorus alone (Placebo Comparator): Effect of phosphorus (500mg) ingestion alone. No meal. Needed to determine the impact of phosphorus alone on DIT
  Interventions: Dietary Supplement: Effect of phosphorus
- high CHO meal alone (Placebo Comparator): Ingestion of placebo tablets with the high carbohydrate meal
  Interventions: Dietary Supplement: Effect of phosphorus
- High CHO meal plus phosphorus (Active Comparator): Effect of phosphorus (500mg) tablets ingestion of DIT of the high carbohydrate meal
  Interventions: Dietary Supplement: Effect of phosphorus
- High protein meal plus phosphorus (Active Comparator): Effect of phosphorus (500mg) tablets ingestion of DIT of the high protein meal
  Interventions: Dietary Supplement: Effect of phosphorus
- High protein meal alone (Placebo Comparator): Ingestion of placebo tablets with the high protein meal
  Interventions: Dietary Supplement: Effect of phosphorus

INTERVENTIONS:
Dietary Supplement: Effect of phosphorus — Ingestion of 500mg of phosphorus ( 4 tablets, each of 125 mg of phosphorus)

SUMMARY:
The study aim at:

Investigating the impact of phosphorus ingestion on DIT of lean and obese subjects consuming high carbohydrate meal.

Investigating the impact of phosphorus ingestion on DIT of lean and obese subjects consuming high protein-low phosphorus meal.

DETAILED DESCRIPTION:
Subject will be advice to take a weight maintenance diet which contains at least 250-300g of carbohydrate per day for the 3 days before each study day and also he/she will be asked to avoid any intense physical activity during the day before the day of the test. Overnight fasted subjects (> 8 hours) will be requested to attend the testing room at around 8:00 am. The he investigators will take the anthropometric measurements (weight, height, waist circumference) and determine blood glucose.

A crossover design study will be used in which each subject will undertake 2 or 3 sessions in a random order over 2 or 3 different days which are separated by a minimum of one week. The difference between the sessions is the ingestion of placebo ( 4 tablets) or phosphorus (4 tablets, each contain 125mgof phosphorus) tablets with the appropriate meal.

Specific Aim 1: The impact of phosphorus ingestion on DIT of lean and obese subjects consuming high carbohydrate meal (Table 1: Meal 1).

This will be divided into two experiments:

Experiment 1.1: The impact of phosphorus ingestion on DIT of lean subjects consuming high carbohydrate meal (16 subjects).

In this experiment, overnight fasted lean subjects (> 8 hours) will be requested to attend the testing room at around 8:00 am. Anthropometric measurements (weight, height, waist circumference) will be taken, rest for 30 min, measure resting energy expenditure (REE) for 30 min, ingest meal with the appropriate supplement and measure postprandial energy expenditure (PEE) for 4 hours (see figure 3). In this experiment, subject will undertake 3 sessions in a random order over 3 different days which are separated by a minimum of one week.

Session 1: Ingestion of phosphorus tablets (4 tablets) alone. No meal. Needed to determine the impact of phosphorus alone on DIT Session 2: Ingestion of phosphorus tablets (4 tablets) with the high carbohydrate meal (table1: Meal 1).

Session 3: Ingestion of placebo tablets (4 tablets) with the high carbohydrate meal (table 1: Meal 1).

Experiment 1.2: The impact of phosphorus ingestion on DIT of lean subjects consuming high carbohydrate meal (16 subjects).

In this experiment, overnight fasted obese subjects (> 8 hours) will be requested to attend the testing room at around 8:00 am. Anthropometric measurements (weight, height, waist circumference) will be taken, rest for 30 min, measure resting REE for 30 min, ingest meal with the appropriate supplement and measure PEE for 4 hours (see figure 3). In this experiment, subject will undertake 3 sessions in a random order over 3 different days which are separated by a minimum of one week.

Session 1: Ingestion of phosphorus tablets (4 tables) alone. No meal. Needed to determine the impact of phosphorus alone on DIT Session 2: Ingestion of phosphorus tablets (4 tables) with the high carbohydrate meal (Table 1:Meal 1).

Session 3: Ingestion of placebo tablets (4 tables) with the high carbohydrate meal (Table 1:Meal 1).

Specific Aim 2: The impact of phosphorus ingestion on DIT of lean and obese subjects consuming high protein-low phosphorus meal (table 1: Meal 2).

This will be divided into two experiments:

Experiment 2.1: The impact of phosphorus ingestion on DIT of lean and obese subjects consuming high protein-low phosphorus meal (16 subjects).

In this experiment, overnight fasted lean subjects (> 8 hours) will be requested to attend the testing room at around 8:00 am. Anthropometric measurements (weight, height, waist circumference) will be taken, rest for 30 min, measure REE for 30 min, ingest meal with the appropriate supplement and measure PEE for 4 hours (see figure 3). In this experiment, subject will undertake 2 sessions in a random order over 2 different days which are separated by a minimum of one week.

Session 1: Ingestion of phosphorus tablets (4 tablets) with the high protein meal (table1: Meal 2).

Session 2: Ingestion of placebo tablets (4 tablets) with the high protein meal (table 1: Meal 2).

Experiment 2.2: The impact of phosphorus ingestion on DIT of lean and obese subjects consuming high protein-low phosphorus meal (16 subjects).

In this experiment, overnight fasted obese subjects (> 8 hours) will be requested to attend the testing room at around 8:00 am. Anthropometric measurements (weight, height, waist circumference) will be taken, rest for 30 min, measure REE for 30 min, ingest meal with the appropriate supplement and measure PEE for 4 hours (see figure 3). Urine sample over the experimental period will be collected. In this experiment, subject will undertake 2 sessions in a random order over 2 different days which are separated by a minimum of one week.

Session 1: Ingestion of phosphorus tablets (4 tablets) with the high protein meal (table1: Meal 2).

Session 2: Ingestion of placebo tablets (4 tablets) with the high protein meal (table 1: Meal 2).

ELIGIBILITY:
Inclusion Criteria:

* lean subjects (BMI between 20 and 25);
* obese (BMI above 30) subjects

Exclusion Criteria:

* Pregnant and lactating women
* Subjects on regular use of medication that affects body weight
* weight loss of 3% or more in the preceding 3 months
* Subjects with kidney disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-07-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in postprandial energy expenditure | 4 hours
  Changes in area under the curve (AUC) of postprandial energy expenditure as measured by determining postprandial the volume oxygen consumption (VO2) and the volume of carbon dioxide production (VCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Obeid, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon